CLINICAL TRIAL: NCT06020911
Title: Clinical and Radiographic Evaluation of Indirect Pulp Capping Using Biodentine and Theracal Light-cured in Primary Molars
Brief Title: Indirect Pulp Capping Using Biodentine and Theracal Light-cured in Primary Molars
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Alaa Abd Elhameed Abd Elghany, Principle investigator Alaa Abd Elhameed Abd Elghany, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-PED-6-21-6
Record Dates: First submitted 2023-08-23; First posted 2023-09-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Pulp Caping; Biodentine; Theracal
MeSH Terms: interventions — tricalcium silicate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biodentine (Active Comparator): 17 primary second molars of 17 children will be capped with Biodentine.
  Interventions: Drug: Biodentine
- Theracal light cured (Active Comparator): 17 primary second molars of 17 children will be capped with Theracal light cured
  Interventions: Drug: Theracal light cured

INTERVENTIONS:
Drug: Biodentine — 17 primary second molars of 17 children will be capped with Biodentine
  Arms: Biodentine
Drug: Theracal light cured — 17 primary second molars of 17 children will be capped with Theracal light cured
  Arms: Theracal light cured

SUMMARY:
this study is aimed to conduct tomographic evaluation of reparative dentin bridges formed after indirect pulp capping with Biodentine and Theracal light cured. The null hypothesis of the study is that there will be no difference in the quantity and quality of reparative dentin formation between the tested materials used for the indirect pulp capping

DETAILED DESCRIPTION:
Many materials have been used in indirect pulp capping for primary dentition. An ideal pulp capping material is to be successful when it is biocompatible, radiopaque, maintain good seal, protect the pulp against bacterial invasion in both long and short run, release sustained amounts of calcium ions, act as reservoir for calcium hydroxide and stimulate reparative dentin formation through inducing the pulp cells to form odontoblasts.

Theracal light cured is a light-cured resin modified calcium silicate (RMCS) used as an indirect pulp capping material. It releases more calcium ions than Mineral trioxide aggregate or dycal inducing reparative dentin and dentin bridge formation.Theracal light cured showed better sealing ability and less microleakage than Mineral trioxide aggregate and Biodentine

ELIGIBILITY:
Inclusion Criteria:

1. Each child has bilateral vital cavitated carious lesions in primary molars.
2. Positive vital pulp testing for both hot and cold response; is determined by ethyl chloride in cold pulp testing and heated gutta percha in hot pulp testing. Pain caused by these tests should not persist after the stimulus is removed.
3. Patient and parent cooperation.
4. Accessible isolation for the operated tooth with rubber dam.
5. primary molars with cavitated carious lesion on either occlusal or proximal surface that extend into the dentin .
6. Availability of remaining dentin thickness over the pulp.
7. Normal lamina dura and periodontal ligaments. 8 Absence of external and internal root resorption.

Exclusion Criteria:

1. Spontaneous pain, or persistent swelling or fistula.
2. Pain with percussion, presence of abscess and pathological mobility.
3. Uncooperative patient.
4. Progression of caries lesion to pulp and pulp exposure.
5. Presence of periapical lesion as abscess, cyst or granuloma.
6. Unhealthy bony tissues.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Thickness of dentin in mm | UP to 9 months postoperatively
  Cone-beam computed tomography(CBCT) scan will be used after placing the capping material once at the start immediately postoperative after restoration and at the end of follow up period after 9 months to evaluate the Thickness of dentin in mm
Radiodenisty in Hounsfield units | UP to 9 months postoperatively
  Cone-beam computed tomography(CBCT) scan will be used after placing the capping material once at the start immediately postoperative after restoration and at the end of follow up period after 9 months to evaluate the Radiodenisty in Hounsfield units
pulp vitality | UP to 9 months postoperatively
  The teeth in each group will be examined clinically after restoration and at the end of the follow up period using vitality tests. Treatment is considered to be successful when pulp remains vital with no signs of pain, no evidence of tooth mobility, normal tooth color, normal gingival health and presence of the restoration intact

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-garbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: after the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author